CLINICAL TRIAL: NCT04329195
Title: ACE Inhibitors or ARBs Discontinuation for Clinical Outcome Risk Reduction in Patients Hospitalized for the Endemic Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Infection: the Randomized ACORES-2 Study
Brief Title: ACE Inhibitors or ARBs Discontinuation in Context of COVID-19 Pandemic
Acronym: ACORES-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recrutment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Hospitalier Pitié-Salpêtrière (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200409
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: History of Cardiovascular Disease Treated With RAS Blockers and With SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Cardiovascular disease; RAS blockers
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: discontinuation of RAS blocker therapy (Experimental): discontinuation of RAS blocker therapy
  Interventions: Drug: 1: discontinuation of RAS blocker therapy
- 2: continuation of RAS blocker therapy (Active Comparator): continuation of RAS blocker therapy
  Interventions: Drug: 2: continuation of RAS blocker therapy

INTERVENTIONS:
Drug: 1: discontinuation of RAS blocker therapy — discontinuation of RAS blocker therapy
  Other Names: discontinuation of RAS blocker therapy
  Arms: 1: discontinuation of RAS blocker therapy
Drug: 2: continuation of RAS blocker therapy — continuation of RAS blocker therapy
  Other Names: continuation of RAS blocker therapy
  Arms: 2: continuation of RAS blocker therapy

SUMMARY:
Since December 2019, a novel coronavirus called SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) has caused an international outbreak of respiratory illness described as COVID-19.

Individuals with a history of cardiovascular disease develop a more severe illness and have higher rates of death.

Because of the potential interaction between RAS blockers and SARS-CoV-2 mechanism of infection, there are ongoing scientific discussions on whether they should be stopped or continued in patients with COVID-19.

It is crucial to determine whether RAS blockers should be discontinued or not in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Chronically treated with RAS blockers (ACE inhibitors or ARBs on the last prescription prior to admission with a treatment duration ≥ 1 month).
* Diagnosis of COVID-19 confirmed by the presence of SARS-CoV-2 on any biological sample with any detection method.
* Patients hospitalized in a non-intensive care unit.
* Pregnancy test at inclusion visit for women of childbearing potential.
* Women of childbearing potential must agree to use adequate contraception according to recommendations related to contraception and pregnancy testing in clinical trials, by Clinical Trial Facilitation Group (CTFG).

Exclusion Criteria:

* Shock requiring vasoactive agents.
* Acute respiratory distress syndrome requiring invasive mechanical ventilation.
* Circulatory assistance.
* History of malignant hypertension according to the definition of the 2018 ESC/ESH guidelines on hypertension.
* Uncontrolled blood pressure despite the use of five antihypertensive drugs.
* History of nephrotic syndrome.
* History of hospitalization for hemorrhagic stroke in the past 3 months.
* RAS blockers therapy previously stopped > 48h.
* No affiliation to the French Health Care System "Sécurité Sociale".
* Inability to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement from day 0 to day 28 (improvement of two points on a seven-category ordinal scale, or live discharge from the hospital, whichever comes first) | from day 0 to day 28 or hospital discharge
  Time to clinical improvement from day 0 to day 28 (improvement of two points on a seven-category ordinal scale, or live discharge from the hospital, whichever comes first)

SECONDARY OUTCOMES:
Primary safety endpoint: major adverse cardiac events defined as the composite of cardiovascular death, myocardial infarction, stroke or acute heart failure at day 28 | at day 28
  Major adverse cardiac events defined as the composite of cardiovascular death, myocardial infarction, stroke or acute heart failure at day 28
Clinical status as assessed with the seven-category ordinal scale on days 7, 14 and 28. | at days 7, 14 and 28
  Clinical status as assessed with the seven-category ordinal scale. The seven-category ordinal scale consisted of the following categories:
  1. not hospitalized with resumption of normal activities
  2. not hospitalized, but unable to resume normal activities
  3. hospitalized, not requiring supplemental oxygen
  4. hospitalized, requiring supplemental oxygen
  5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both
  6. hospitalized, requiring ECMO, invasive mechanical ventilation, or both
  7. death.
Number of days alive free of oxygen. | from day 0 to day 28 or hospital discharge
  Number of days alive free of oxygen.
Number of days alive outside hospital until day28 | at day28
  Number of days alive outside hospital
Number of days alive free of intensive-care unit (ICU) admission or mechanical Ventilation (invasive or non-invasive) until day28 | at day28
  Ventilation (invasive or non-invasive)
Number of days alive free of mechanical ventilation (invasive or non-invasive) until day28 | at day28
  Number of days alive free of mechanical ventilation (invasive or non-invasive)
Number of days alive free of ICU admission until day28 | at day28
  Number of days alive free of ICU admission
Rate of all-cause mortality at day 28 | at day 28
  Rate of all-cause mortality
Rate of cardiovascular death at day 28 | at day 28
  Rate of cardiovascular death
Number of days alive free of acute kidney injury until hospital discharge | at day 28 to hospital discharge
  Number of days alive free of acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, MD, PhD, Principal Investigator — Institut Cardiologie - Pitié Salpêtrière(APHP) / ACTION Study Group / Univ. Paris 6 (UPMC) - INSERM UMRS 1166
Locations (1):
- Cardiologie, Groupe Hospitalier Pitié-Salpêtrière, Paris, France